CLINICAL TRIAL: NCT02926066
Title: A Clinical Trial for Treatment of Aromatic L-amino Acid Decarboxylase (AADC) Deficiency Using AAV2-hAADC - An Expansion (NTUH-AADC-011)
Brief Title: A Clinical Trial for Treatment of Aromatic L-amino Acid Decarboxylase (AADC) Deficiency Using AAV2-hAADC - An Expansion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201511036MIND
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2022-11

CONDITIONS: Aromatic Amino Acid Decarboxylase Deficiency
Keywords: Aromatic L-amino acid decarboxylase (AADC)
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AAV2-hAADC (Experimental): Dosage form: Aqueous solution Dose(s): 2.37x10^11 vg/case(High dose) Dosing schedule: Intracerebral infusion, single dose Mechanism of action (if known): supplement a gene defect
  Dosage form: Aqueous solution Dose(s): 1.81x10^11 vg/case(Standard dose) Dosing schedule: Intracerebral infusion, single dose Mechanism of action (if known): supplement a gene defect
  Interventions: Drug: AAV2-hAADC

INTERVENTIONS:
Drug: AAV2-hAADC — Dosage form: Aqueous solution Dose(s): 2.37x10^11 vg/case(High dose) Dosing schedule: Intracerebral infusion, single dose Mechanism of action (if known): supplement a gene defect
  Dosage form: Aqueous solution Dose(s): 1.81x10^11 vg/case(Standard dose) Dosing schedule: Intracerebral infusion, single dose Mechanism of action (if known): supplement a gene defect

SUMMARY:
This clinical trial expansion is to offer patients, who are not enrolled into the Phase I/II trial, a chance of treatment, to provide the experience in this gene therapy, and to increase the dose slightly.

DETAILED DESCRIPTION:
AAV2-hAADC will be made by a GMP laboratory. An MRI will be performed to define the brain structure, and then metal nails will be fixed on the skull and a CT will be performed. The two images will be confined and the direction and depth of infusion will be determined. During the surgery, a stereotactic device will be implanted on both sides of the brain on a bur hole. Each putamen will be injected for two times. If there is no complication from the surgery, the patients will enter the follow up period.

In Cohort 1, subjects for high dose (2.37x10^11 vg) will be enrolled via sequential enrollment with an observation for 2 months or even longer. Only after a subject passing peak dyskinesia, which is indicated by a reduced drug dose required for alleviation of dyskinesia, or improved food intake, and being verified by Safety Committee, treatment for the next patient with high dose can be proceeded.

In Cohort 2, in order to be compared with Phase I/II (n=10), 4 patients will be treated in Cohort 2 and all of them will use the high dose (2.37x10^11 vg). Patients older than 3 (no more than 2 patients) years of age will be enrolled via sequential enrollment with an observation for 2 months or longer. Only after a subject passing peak dyskinesia, which is indicated by a reduced drug dose required for alleviation of dyskinesia, or improved food intake, which has been verified by the Safety Committee can the treatment at a high dose begin in the next patient older than 3.

ELIGIBILITY:
Inclusion Criteria:

1. With a confirmed diagnosis of AADC, including cerebrospinal fluid analysis to show reduced levels of neurotransmitter metabolites, HVA and 5-HIAA, and higher L-Dopa, or with more than one mutation within AADC gene, etc.
2. Classical clinical characteristics of AADC deficiency, such as oculogyric crises, hypotonia and developmental retardation.
3. The child patient has to be over 2 years old or a thickness of skull enough for surgery.
4. The child patient has to be under 6 years old (72 months) before being treated with study drugs.
5. Participating patients must cooperate completely for all evaluations and examinations before, during and after the whole trial.
6. Parents or guardians must sign to agree on this informed consent.

Exclusion criteria:

1. Significant brain structure abnormality determined by the physician.
2. Patients with any health or neurological doubts that may increase the risk of surgery cannot join this trial. PI has the right to evaluate the feasibility of subjects for this trial based on his/her health condition.
3. Patients with anti-AAV2 neutralizing antibody titer over 1,200 folds or an ELISA OD over 1 cannot be recruited into this trial.
4. Subjects participating in this trial cannot take any medications that may affect this clinical trial, which do not apply to those drugs used at specified duration as mentioned in this protocol.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of therapeutic effect | 13 months
  1. At one year post-surgery, neurotransmitter metabolites (HVA or HIAA) increased in the CSF (compared to the pre-surgery (Baseline) level).
  2. At one year post-surgery, PDMS-II score is higher than that at pre-surgery (Baseline), with an improvement over 10 points.

SECONDARY OUTCOMES:
Evaluation for the treatment safety | 13 months
  1. The absence of intracranial bleeding, which requires surgical management, after the surgery
  2. Craniotomy-induced CSF exudation
  3. The severity of post-surgery dyskinesia (if feeding is affected and then nasogastric tube is required)
  4. Incidence of other severe adverse events (information of adverse events of all kinds and severities will be collected, including treatment-emergent adverse events).
Evaluation of secondary therapeutic effects | 13 months
  1. Weight gain
  2. Increased signal intensity of dopamine in putamen during PET imaging
  3. Increased score in other development evaluations
Exploratory endpoint | 13 months
  1. The correlation between AAV2 antibody titer and therapeutic effect
  2. The correlation between subject's age and therapeutic effect

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, MD.,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tai CH, Lee NC, Chien YH, Byrne BJ, Muramatsu SI, Tseng SH, Hwu WL. Long-term efficacy and safety of eladocagene exuparvovec in patients with AADC deficiency. Mol Ther. 2022 Feb 2;30(2):509-518. doi: 10.1016/j.ymthe.2021.11.005. Epub 2021 Nov 8. PMID 34763085